CLINICAL TRIAL: NCT04001049
Title: Glycemic Variability: Prognostic Impact on Acute Ischemic Stroke and Impact of the Corrective Treatment for Hyperglycemia.
Brief Title: Glycemic Variability: Prognostic Impact on Acute Ischemic Stroke
Acronym: GLIAS-III
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: GLIAS-III
Record Dates: First submitted 2019-05-22; First posted 2019-06-27 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Brain Ischemia; Hyperglycemia; Glycemic Variability
MeSH Terms: conditions — Brain Ischemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter observational clinical study in patients with acute ischemic stroke. The main objective is to evaluate the impact of glycemic variability (GV) on stroke outcome (mortality, functional recovery) of patients with acute ischemic stroke. Glycemic variability will be assessed using a subcutaneous device for continuous glycaemia motorization during 96 hours; also capillar glycaemia will be measured every 6 hours.

DETAILED DESCRIPTION:
10 different hospitals in Spain will participate in this study, recruiting a total of 340 patients. Once the informed consent form is signed, the subcutaneous device for continuous glycaemia motorization will be implanted and demographic, comorbidities and treatments of every patient will be registered. During the first 96 hours, capillar glycaemia, NIHSS scale, HbA1C levels, cerebral recanalization treatment and glycaemia correcting treatments will also be reported. In the following days (7, 30 and 90 days after stroke) modified Rankin Scale, NIHSS scale and stroke secondary prevention treatments will be evaluated. At day 90, a new measure of HbA1C will be done.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Inclusion less than 24 hours from ischemic stroke
* Functional independence prior to stroke
* Signed informed consent

Exclusion Criteria:

* Transient cerebral ischemia
* Prevision of need to perform a magnetic resonance within the first 96 hours from inclusion
* Concomitant severe or deadly disease that may interfere with study follow-up during 3 months from stroke
* Current drug or alcohol abuse that may interfere with study follow-up
* Participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years old presenting with acute ischemic stroke of less than 24 hours of evolution
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic variation impact in mortality of patients with acute ischemic stroke | 3 months from stroke
  Intrahospital mortality
Glycemic variation impact in functional status of patients with acute ischemic stroke | 3 months from stroke
  Modified Rankin Scale. This scale measures degree of disability/dependence after a stroke.
  0- No symptoms
  1. No significant disability despite symptoms; able to perform all usual duties and activities.
  2. Slight disability; unable to perform all previous activities but able to look after own affairs without assistance.
  3. Moderate disability; requires some help but able to walk without assistance.
  4. Moderate severe disability; unable to walk without assistance an unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requires constant nursing care and attention.
  6. Death

SECONDARY OUTCOMES:
Impact of glycemic variation in mortality in diabetic patients with acute ischemic stroke. | 3 months from stroke
  Intrahospital mortality
Impact of glycemic variation in functional status in diabetic patients with acute ischemic stroke. | 3 months from stroke
  Modified Rankin Scale. This scale measures degree of disability/dependence after a stroke.
  0- No symptoms
  1. No significant disability despite symptoms; able to perform all usual duties and activities.
  2. Slight disability; unable to perform all previous activities but able to look after own affairs without assistance.
  3. Moderate disability; requires some help but able to walk without assistance.
  4. Moderate severe disability; unable to walk without assistance an unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requires constant nursing care and attention.
  6. Death

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Fuentes Gimeno, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fuentes B, Pastor-Yborra S, Gutierrez-Zuniga R, Gonzalez-Perez de Villar N, de Celis E, Rodriguez-Pardo J, Gomez-de Frutos MC, Laso-Garcia F, Gutierrez-Fernandez M, Ortega-Casarrubios M, Soto A, Lopez-Fernandez M, Santamaria M, Diez-Gonzalez N, Freijo MM, Zandio B, Delgado-Mederos R, Calleja A, Portilla-Cuenca JC, Lisbona A, Otero-Ortega L, Diez-Tejedor E. Glycemic variability: prognostic impact on acute ischemic stroke and the impact of corrective treatment for hyperglycemia. The GLIAS-III translational study. J Transl Med. 2020 Nov 4;18(1):414. doi: 10.1186/s12967-020-02586-4. PMID 33148277